CLINICAL TRIAL: NCT00002721
Title: A PHASE I TRIAL OF ESTRAMUSTINE PHOSPHATE AND DOXORUBICIN IN HORMONE REFRACTORY METASTATIC PROSTATE CANCER
Brief Title: Doxorubicin Plus Estramustine in Treating Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNM-2394C; CDR0000064574 (Registry Identifier: PDQ (Physician Data Query)); NCI-V96-0816
Record Dates: First submitted 1999-11-01; First posted 2004-05-26 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Doxorubicin; Estramustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prostate cancer patients (Experimental): Prostate cancer patients that have not responded to hormon therapy
  Interventions: Drug: doxorubicin hydrochloride; Drug: estramustine phosphate sodium; Procedure: drug resistance inhibition treatment

INTERVENTIONS:
Drug: doxorubicin hydrochloride
Drug: estramustine phosphate sodium
Procedure: drug resistance inhibition treatment

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of doxorubicin plus estramustine in treating patients with metastatic recurrent prostate cancer that does not respond to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the maximum tolerated dose of weekly intravenous doxorubicin (DOX) that can be given in combination with oral estramustine (EM) in patients with metastatic prostate cancer refractory to treatment with hormonal agents. II. Assess the frequency of expression of the multidrug resistance phenotype in biopsy specimens from these patients. III. Assess the response to DOX/EM in these patients.

OUTLINE: 2-Drug Combination Chemotherapy. Doxorubicin, DOX, NSC-123127; Estramustine, EM, NSC-89199.

PROJECTED ACCRUAL: Three to 18 patients will be entered.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Biopsy proven metastatic prostate cancer Biopsy requirement waived at principal investigator's discretion if new disease site technically inaccessible and PSA elevated Recurrent disease following orchiectomy, estrogen, or gonadotropin-releasing hormone agonist therapy If previously irradiated: Progressive disease outside prior radiotherapy field required No brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 1.5 mg/dL ALT/AST less than 3 times greater than normal Renal: Not specified Cardiovascular: Left ventricular ejection fraction at least 45% No NYHA class III/IV status No unstable angina Other: No Crohn's disease, ulcerative colitis, or other inflammatory bowel syndrome

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior doxorubicin or estramustine Endocrine therapy: See Disease Characteristics At least 30 days since flutamide Estrogen or gonadotropin-releasing hormone agonists discontinued prior to treatment Radiotherapy: At least 6 weeks since radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 1995-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Respond to therapy | six months

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Y. Smith, MD, Study Chair — University of New Mexico Cancer Center
Locations (1):
- University of New Mexico Cancer Research & Treatment Center, Albuquerque, New Mexico, United States